CLINICAL TRIAL: NCT00356070
Title: Treatment of Prisoners With Attention Deficit Hyperactive Disorder in Trondheim Prison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AH 4.2005.147
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder, treatment,; Strattera,; rehabilitation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Strattera

SUMMARY:
The treatment of ADHD in jail will help the prisoners in their rehabilitation process

DETAILED DESCRIPTION:
Prisoners with ADHD will be offered treatment with Stratera, and we wanted to study their use of the prisons rehabilitation offers as school, programs and work training before and after treatment with Stratera.

ELIGIBILITY:
Inclusion Criteria:

All prisoners that fullfill the diagnostic criterias for ADHD -

Exclusion Criteria:

All other prisoners -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-01 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The symptoms of Attention Deficit Hyperactive Disorders and the prisoners use of the prisons rehabilitation services before and after treatment will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Roger Almvik, md phd, Principal Investigator — St. Olavs Hospital, Departement of forensic psychiatry, Brøset
Locations (1):
- St. Olavs Hospital. Departement for forensic psyciatry, Brøset., Trondheim, Norway